CLINICAL TRIAL: NCT05340153
Title: Efficacy and Safety of Artemether-Lumefantrine and Dihydroartemisinin-Piperaquine for the Treatment of Uncomplicated Plasmodium Falciparum Malaria Among Children in the North Region of Cameroon
Brief Title: Efficacy and Safety of Artemether-Lumefantrine and Dihydroartemisinin-Piperaquine in Cameroon
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Yaounde 1 (Other)
Collaborators: Biotechnology Center (BTC), University of Yaounde I, Cameroon (Unknown); National Malaria Control Program (NMCP), Cameroon (Unknown); Association Camerounaise pour le Marketing Social (ACMS), Cameroon (Unknown); Impact Malaria, Cameroon (Unknown)
Responsible Party: Principal Investigator, Professor Wilfred Fon Mbacham, Principal Investigator, Professor of Public Health Biotechnology, University of Yaounde 1
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AAAL002/PMI/CMR
Record Dates: First submitted 2022-04-11; First posted 2022-04-22 (Actual); Last update posted 2022-04-22 (Actual); Status verified 2022-04

CONDITIONS: Malaria
Keywords: Plasmodium falciparum; Malaria; Artemether-lumefantrine; Dihydroartemisinin-piperaquine; Cameroon
MeSH Terms: conditions — Malaria; Malaria, Falciparum | interventions — Artemether, Lumefantrine Drug Combination

STUDY DESIGN:
Intervention Model Description: Eligible children for whom parent/guardian authorization and assent are obtained will be randomized to receive either artemether-lumefantrine (group A) or dihydroartemisinin-piperaquine (group B) in the ratio 1:1
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Artemether-lumefantrine (Active Comparator): Drug: Artemether-lumefantrine drug combination Artemether-lumefantrine is formulated as tablets and will be provided in blister packs. Each tablet contains 20 mg artemether and 120 mg lumefantrine. Every pack has a picture showing how the drug should be given and contains a blister of 12 tablets. It will be administered each day as one, two or three tablets depending on the weight of the child.
  Interventions: Drug: Artemether-Lumefantrine Drug Combination
- Dihydroartemisinin-piperaquine (Experimental): Drug: Dihydroartemisinin-piperaquine drug combination Dihydroartemisinin-piperaquine is formulated as tablets and will be provided in blister packs. Each tablet contains 40 mg dihydroartemisinin and 320 mg piperaquine. Every pack has a picture showing how the drug should be given and contains a blister of 6 tablets and given each day as half, one, two or three tablets depending on the weight of the child.
  Interventions: Drug: Dihydroartemisinin-Piperaquine drug combination

INTERVENTIONS:
Drug: Artemether-Lumefantrine Drug Combination — Artemether-lumefantrine is formulated as tablets and will be provided in blister packs. Each tablet contains 20 mg artemether and 120 mg lumefantrine. Every pack has a picture showing how the drug should be given and contains 1 blister of 12 tablets. It will be administered each day as two, four, six or eight tablets depending on the weight of the child.
  Other Names: Coartem dispersible
  Arms: Artemether-lumefantrine
Drug: Dihydroartemisinin-Piperaquine drug combination — Dihydroartemisinin-piperaquine is a formulated as tablets and will be provided in blister packs. Each tablet contains 40 mg dihydroartemisinin and 320 mg piperaquine. Every pack has a picture showing how the drug should be given and contains 1 blister of 6 tablets. It will be given each day as a half, one, two or three tablets depending on the weight of the child.
  Other Names: D-ARTEPP dispersible
  Arms: Dihydroartemisinin-piperaquine

SUMMARY:
Malaria is an infectious disease transmitted by the bite of an infected female anopheles mosquito. The most vulnerable group that bears the highest disease burden includes children less than five years and pregnant women. Artemether-lumefantrine (AL) has been used for the treatment of uncomplicated Plasmodium falciparum in Cameroon since 2006. In 2020, the government of Cameroon also adopted the use of dihydroartemisinin-piperaquine (DHA-PPQ) as one of the first line drugs for the treatment of malaria. Globally, several studies among children have reported high efficacy and safety of artemisinin-based combination therapies (ACTs). However, there is paucity of data to support the continuous use of AL and DHA-PPQ in Cameroon. The main objective of this study is to assess the efficacy and safety of artemether-lumefantrine (AL) and dihydroartemisinin-piperaquine (DHA-PPQ) uncomplicated P. falciparum malaria in the North Region of Cameroon. A randomized, open-label, controlled clinical trial comparing artemether-lumefantrine (AL) and dihydroartemisinin-piperaquine (DHA-PPQ) will be carried out from 11th April to 31st December, 2022 at two hospitals in the North Region of Cameroon. The study participants shall include febrile patients aged 6 months to 10 years with confirmed uncomplicated P. falciparum infection. Eligible children for whom parent/guardian assents are obtained will be randomized to receive either artemether-lumefantrine (group A) or dihydroartemisinin-piperaquine (group B) in the ratio 1:1. A minimum sample of 76 patients will be required for the study. With a 20 % increase to allow loss to follow-up and withdrawals during the 28-days (AL) or 42-days (DHA-PPQ) follow-up period, 92 patients will be enrolled into each of the two study arms. The study will recruit a total of 184 patients. However, since 2 study sites will be involved, a minimum of 92 (46 per drug arm) participants shall be enrolled per site. Drug intake will be done under strict supervision on days 0, 1 and 2. Follow-up visits will be performed on days 3, 7, 14, 21, 28, 35 and 42 to evaluate clinical and parasitological resolution of their malaria episode as well as adverse events. Polymerase chain reaction (PCR) of Plasmodium falciparum merozoite surface proteins 1 and 2 (Pfmsp1, Pfmsp2), glutamate-rich protein (Pfglurp) and microsatellites will be used to differentiate between recrudescence and new infection.

DETAILED DESCRIPTION:
Brief title: Efficacy and Safety of Artemether-Lumefantrine (AL) and Dihydroartemisinin-Piperaquine (DHA-PPQ) in Cameroon

Official title: Efficacy and Safety of Artemether-Lumefantrine and Dihydroartemisinin-Piperaquine for the treatment of uncomplicated Plasmodium falciparum malaria among children in the North Region of Cameroon

Purpose: To assess the efficacy and safety of artemether-lumefantrine (AL) and dihydroartemisinin-piperaquine (DHA-PPQ) for the treatment of uncomplicated P. falciparum malaria among children 6 to 120 months at District Hospital Figuil and District Hospital Guider in the North Region of Cameroon.

Background: Malaria is an infectious disease transmitted by the bite of an infected female anopheles mosquito. The most vulnerable group includes children less than five years and pregnant women. artemether-lumefantrine (AL) has been used for the treatment of uncomplicated Plasmodium falciparum in Cameroon since 2006. In 2020, the government of Cameroon also adopted the use of dihydroartemisinin-piperaquine (DHA-PPQ) as one of the first line drugs for the treatment of malaria. Globally, several studies among children have reported high efficacy and safety of artemisinin-based combination therapies (ACTs). However, there is paucity of data to support the continuous use of AL and DHA-PPQ in Cameroon.

Objective: To assess the efficacy and safety of artemether-lumefantrine (AL) and dihydroartemisinin-piperaquine (DHA-PPQ) for the treatment of uncomplicated P. falciparum malaria among children 6 to 120 months at District Hospital Figuil and District Hospital Guider in the North Region of Cameroon.

Study sites: District Hospital Guider and District Hospital Figuil in the North Region of Cameroon.

Study period: 11th April to 31st December 2022.

Study design: This surveillance study is a two-arm, open-label, randomized controlled clinical trial.

Patient population: Febrile patients aged 6 months to 10 years, with confirmed uncomplicated P. falciparum infection. Eligible children for whom parent/guardian informed consents are obtained will be randomized to receive either artemether-lumefantrine (group A) or dihydroartemisinin-piperaquine (group B) in the ratio 1:1.

Sample size: A minimum sample of 76 patients will be required for the study. With a 20 % increase to allow for loss to follow-up and withdrawals during the 28-days and 42-days follow-up period, 92 patients will be enrolled for each of the two study arms. The study will recruit a total of 184 patients. At least 46 participants shall be enrolled into each drug arm of at the two sites.

Treatment (s) and follow-up: Drug intake will be done under strict supervision on days 0, 1 and 2. Follow-up visits will be performed on days 3, 7, 14, 21, 28 (AL), 35 and 42 (DHA-PPQ) to evaluate clinical and parasitological resolution of their malaria episode as well as adverse events. Polymerase chain reaction (PCR) of Plasmodium falciparum merozoite surface proteins 1 and 2 (Pfmsp1, Pfmsp2), glutamate-rich protein (Pfglurp) and microsatellites will be used to differentiate between recrudescence and new infection.

Classification of treatment outcomes: Classification of treatment outcomes will be done based on the WHO 2009 guidelines: treatment failure (Early Treatment Failure-ETF, Late Clinical failure-LCF and Late Parasitological Failure-LPF) and treatment success (Adequate Clinical and Parasitological Response-ACPR).

ELIGIBILITY:
Inclusion Criteria:

* Children of either gender, aged 6 months to 10 years will be recruited.
* Uncomplicated P. falciparum malaria confirmed by microscopy using Giemsa-stained thick film with an asexual parasite density within the range of 1000 to 200000 parasites/μl.
* Presenting with fever (axillary temperature ≥ 37.5 ºC) or having a history of fever in the preceding 24 hours.
* Able to ingest tablets orally (either suspended in water or uncrushed with food).
* Willing to participate in the study with written informed consent from parent/guardian.
* Willing and able to attend the clinic on stipulated regular follow-up visits.

Exclusion Criteria:

* Mixed or mono-infection with another Plasmodium species detected by microscopy.
* Children who are currently suffering or had the following within the last 2 months: tuberculosis, HIV, schistosomiasis, diabetes mellitus, cardiovascular disease, gout, rheumatoid arthritis, underlying chronic hepatic or renal disease, hypoglycemia, jaundice, respiratory distress, and other inflammatory-related diseases.
* Signs/symptoms indicating severe/complicated malaria" according to WHO criteria (WHO definition) such as:

  1. Not able to drink or breastfeed.
  2. Persistent vomiting (>2 episodes within the previous 24 hours).
  3. Convulsions (>1 episode within the previous 24 hours).
  4. Lethargic/unconscious.
  5. Severe anemia (hemoglobin < 5 g/dl).
* Serious gastrointestinal disease.
* Presence of severe malnutrition defined as a child aged between 6-60 months whose weight-for-height is below -3 z-score (W/H < 70%) or has symmetrical edema involving at least the feet or has a mid-upper arm circumference <115 mm).
* Regular medication, which may interfere with antimalarial pharmacokinetics.
* History of hypersensitivity reactions or contraindications to any of the medicine (s) being tested or used as alternative treatment (s).
* Individuals who have taken part in anti-malarial efficacy and safety studies in the last 3 months.
* Participants who have taken antimalarial drugs within the last one month.

Ages: 6 Months to 120 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 184 (Estimated)
Dates: Start 2022-04-11 (Estimated); Primary Completion 2022-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
The number of participants with treatment success and adverse events following treatment with AL and DHA-PPQ in children infected with uncomplicated P. falciparum malaria. | 10 months
  Eligible children for whom parent/guardian informed consents are obtained will be randomized to receive either artemether-lumefantrine (group A) or dihydroartemisinin-piperaquine (group B) in the ratio of 1:1.

SECONDARY OUTCOMES:
The proportion of patients with early treatment failure, late clinical failure, late parasitological failure or an adequate clinical and parasitological response as indicators of efficacy according to the WHO 2009 guidelines. | 10 months
  Eligible children for whom parent/guardian informed consents are obtained will be randomized to receive either artemether-lumefantrine (group A) or dihydroartemisinin-piperaquine (group B) in the ratio of 1:1.
  Recrudescence will be distinguished from re-infection by polymerase chain reaction (PCR) analysis.
The number of participants with treatment-related adverse events as assessed by CTCAE v4.0. | 10 months
  Eligible children for whom parent/guardian informed consents are obtained will be randomized to receive either artemether-lumefantrine (group A) or dihydroartemisinin-piperaquine (group B) in the ratio of 1:1.
The number of children with single nucleotide polymorphisms of P. falciparum genes responsible for resistance to AL and DHA-PPQ. | 10 months
  Pre-treatment and recrudescence/reinfection samples during follow-up shall be used to characterize the molecular markers of Plasmodium falciparum chloroquine resistant transporter(Pfcrt), Plasmodium falciparum multi-drug resistant 1 (Pfmdr1), and Plasmodium falciparum K13 (Pfk13) propeller domain conferring resistance to artemisinins or partner drugs.
The number of children with single nucleotide polymorphisms of P. falciparum histidine-rich protein 2 and 3 genes. | 10 months
  Pre-treatment shall be used to detect single nucleotide polymorphisms present in Plasmodium falciparum histidine-rich protein 2 and 3 genes.

CONTACTS AND LOCATIONS:
Overall Officials: Wilfred Fon Mbacham, PhD, Principal Investigator — University of Yaounde I

IPD SHARING:
Plan to Share IPD: Yes
Research findings will be communicated to the scientific community and policymakers. This will be done through public engagements and publications in peer-review journals.
Supporting Information: Study Protocol, CSR
Time Frame: 31st December 2022 for at least 10 years
Access Criteria: Not available for now